CLINICAL TRIAL: NCT06326385
Title: Development and Validation of Predictive Models for Sepsis Risk in Patients With Intracerebral Hemorrhage in Intensive Care Units Based on Machine Learning: A Retrospective Cohort Study
Brief Title: Machine Learning Predictive Models for Sepsis Risk in ICU Patients With Intracerebral Hemorrhage
Status: Not yet recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 53244021
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Intracerebral Hemorrhage; Sepsis
MeSH Terms: conditions — Cerebral Hemorrhage; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intracerebral hemorrhage
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Patients with intracerebral hemorrhage (ICH) in the intensive care unit (ICU) are at heightened risk of developing sepsis, significantly increasing mortality and healthcare burden. Currently, there is a lack of effective tools for the early prediction of sepsis in ICH patients within the ICU. This study aims to develop a reliable predictive model using machine learning techniques to assist clinicians in the early identification of patients at high risk and to facilitate timely intervention.

The Medical Information Mart for Intensive Care (MIMIC) IV database (version 2.2) is an international online repository for critical care expertise. This database contains patient-related information collected from the ICUs of Beth Israel Deaconess Medical Center between 2008 and 2019. It includes a vast dataset of 299,712 hospital admissions and 73,181 intensive care unit patients.

The eICU Collaborative Research Database (eICU-CRD) comprises data from over 200,000 ICU admissions for 139,367 unique patients across 208 US hospitals between 2014 and 2015, providing a valuable resource for critical care research.

This study aims to establish and validate multiple machine learning models to predict the onset of sepsis in ICU patients with ICH and to identify the model with the optimal predictive performance.

DETAILED DESCRIPTION:
* Data Collection: This study utilized two public databases. The model leveraged clinical data obtained from the Medical Information Mart for Intensive Care (MIMIC) IV database (version 2.2) and selected corresponding patients for external validation from the eICU Collaborative Research Database (eICU-CRD). Data on ICH patients were extracted from the MIMIC IV public database, including baseline characteristics, clinical parameters, therapeutic interventions, and outcomes. The data were randomly divided into two groups, with 70% serving as the training set and 30% as the validation set.
* Model Development: Feature selection was performed using Lasso regression to construct various machine learning models (such as Random Forest, Logistic Regression, and Neural Networks).
* Model Validation: In addition to the internal validation set, external validation was also conducted on the eICU database to test the model's generalizability.
* Statistical Analysis: The predictive performance of the model was evaluated using metrics including the area under the ROC curve (AUC), sensitivity, and specificity.
* Clinical Applicability Assessment: The clinical utility of the model was assessed using Decision Curve Analysis (DCA).

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed with primary intracerebral hemorrhage by ICD-9/10 coding.
* 2. Aged 19-89 years old.

Exclusion Criteria:

* 1. Patients admitted to the hospital but not to the ICU.
* 2. Patients with missing follow-up data or incomplete variables.
* 3. Patients with a hospital stay exceeding one month.

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All diagnoses in the MIMIC-IV and the eICU-CRD databases were identified based on the International Classification of Diseases, Ninth Revision (ICD-9), and ICD-10 codes. For the analysis, patients diagnosed with ICH were included. Sepsis was defined according to the Third International Consensus Definition of Sepsis and Septic Shock (Sepsis-3), which considers patients with suspected infection and a Sequential Organ Failure Assessment (SOFA) score ≥2 as septic.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of sepsis | within 30 days of admission
  Occurrence of sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- Le Zhang, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
In the paper